CLINICAL TRIAL: NCT02987335
Title: Metabolic Characteristics of Lean Diabetes in Rural and Semi-urban India and in the United States
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Meredith Hawkins, Professor of Medicine, Albert Einstein College of Medicine
Other Study IDs: 2013-2191; R01DK079974 (NIH); R01DK069861 (NIH)
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Results first posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Malnutrition; Diabetes; Diabetes
Keywords: Diabetes; Malnutrition
MeSH Terms: conditions — Malnutrition; Diabetes Mellitus | interventions — Constriction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, Fat Biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Lean Diabetes Subjects: N=20 subjects with BMI 16-22.5 kg/m2, with a history of low birth weight and malnutrition documented on at least one occasion. Will undergo pancreatic clamp.
  Interventions: Drug: Pancreatic Clamp
- Type 2 Diabetes Mellitus Subjects: N=13 subjects with BMI 22.5-27 kg/m2. Will undergo pancreatic clamp
  Interventions: Drug: Pancreatic Clamp
- Type 1 Diabetes Mellitus Subjects: N=15 subjects with BMI 16-22.5 kg/m2. Will undergo pancreatic clamp
  Interventions: Drug: Pancreatic Clamp
- Lean Nondiabetic Subjects: N=16 nondiabetic with BMI 16-22.5 kg/m2 subjects 19-45 years of age and in general good health, taking no medications, with normal glucose tolerance and no family history of diabetes. These subjects will be similar in age, ethnicity and BMI with the lean DM group, and will be recruited through various means of community outreach, including notices in shops and newspapers. Will undergo pancreatic clamp
- Obese Nondiabetic Subjects: N=9 nondiabetic with BMI 16-22.5 kg/m2 subjects 19-45 years of age and in general good health, taking no medications, with normal glucose tolerance and no family history of diabetes. These subjects will be similar in age, ethnicity and BMI with the Type 2 diabetes Mellitus group, and will be recruited through various means of community outreach, including notices in shops and newspapers. Will undergo pancreatic clamp

INTERVENTIONS:
Drug: Pancreatic Clamp — We are not performing any interventions; we are only characterizing participants using tests. The hormones that we are administering are not a treatment but are typically used in context of routine care.
  Other Names: Clamp
  Groups: Lean Diabetes Subjects; Type 1 Diabetes Mellitus Subjects; Type 2 Diabetes Mellitus Subjects

SUMMARY:
This purpose of this study is to define the metabolic characteristics of individuals with Lean Diabetes. We aim to determine whether differences in body composition, including any differences in lipid (fat) deposition, exist compared to individuals with either known forms of diabetes (eg, type 1 and type 2), or individuals without diabetes. Diabetes affects the ability of the body to process glucose (sugar). Therefore, we also plan to investigate the ability of the hormone insulin to regulate changes in glucose in these individuals. Developing a greater understanding of the features of this condition could have tremendous therapeutic benefit for these individuals.

DETAILED DESCRIPTION:
India has the world's highest prevalence of diabetes, expected to rise to 80 million by 2030. This includes many patients with Lean Diabetes, which is a form of diabetes identified clinically by early onset, high insulin requirements, absence of other pancreatic disease, and low body mass index (typically ≤17 kg/m2) at presentation. Despite its prevalence, Lean Diabetes remains a relatively unknown disease that stirs conflicting opinions regarding its classification, diagnostic criteria, and pathogenesis.

In this study, the investigators will study individuals meeting the criteria for Lean Diabetes, Type 1 diabetes, Type 2 diabetes, and two group of participants without diabetes using a procedure called a "pancreatic clamp" study. During the clamp procedure, glucose (a sugar) and insulin (a hormone produced in the pancreas that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism. Endogenous glucose production (a measure of the body's production of sugar) will also be measured. Participants will also have a fat biopsy, and will be given a mixed meal challenge which is a test that detects hyperglycemia and glucose intolerance.

The overall goal of this study is to define the metabolic characteristics of individuals with Lean Diabetes and to determine which differences exist compared to individuals with other known forms of diabetes or individuals without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-45 yr
* Diabetes duration at least one year (for the diabetes groups)
* BMI range: 16-22.5 kg/m2 (individuals with lean and type 1 diabetes and non-diabetic controls); 22.5-27 kg/m2 in individuals with type 2 diabetes
* Negative GAD antibodies
* Present (>1.0pmol/l) C-peptide response to Sustacal challenge
* Stable and moderate-to-poor glycemic control (HbA1c greater than 8%)
* Able and willing to provide informed consent.

Exclusion Criteria:

* Mentally disabled persons
* Major psychiatric disorder on medication (excluding successfully treated depression)
* HIV/AIDS
* History of any cancer
* Alcohol or substance abuse or toxin exposure which could be associated with neuropathy
* Cushing's syndrome
* Pregnancy or breast-feeding
* Untreated or uncontrolled hypertension
* Any Chronic illness requiring medication
* History of bleeding disorder or with a prolonged PT or PTT
* Renal disease
* Liver impairment
* Prisoners

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from the community and outpatient practices in India. Diabetes subjects must meet the following criteria: Age 19-45 years, diabetes duration at least one year, negative GAD antibodies, >1.0pmol/l C-peptide response to meal, stable and moderate glycemic control (HbA1c 8-11%), no pancreatic calcification, and not suffering from complications. Subjects will be otherwise in good health. Non diabetic subjects (ND): BMI 16-22.5kg/m2 (lean ND) and BMI 24.5-29.5 (obese ND), Age 19-45 years and in general good health, and no family diabetic history. Subjects will be recruited through various means of community outreach.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Hawkins, Principal Investigator — Albert Einstein College of Medicine

RESULTS

PARTICIPANT FLOW:
Groups:
- Lean Diabetes Subjects: N=20 subjects with BMI 16-19.5 kg/m2, with a history of low birth weight and malnutrition documented on at least one occasion. Will undergo pancreatic clamp.
  Pancreatic Clamp: We are not performing any interventions; we are only characterizing participants using tests. The hormones that we are administering are not a treatment but are typically used in context of routine care.
- Lean Nondiabetic Subjects: N=16 nondiabetic with BMI 16-22.5 kg/m2 subjects 19-45 years of age and in general good health, taking no medications, with normal glucose tolerance and no family history of diabetes. These subjects will be similar in age, ethnicity and BMI with the lean DM group, and will be recruited through various means of community outreach, including notices in shops and newspapers. Will undergo pancreatic clamp
  Pancreatic Clamp: We are not performing any interventions; we are only characterizing participants using tests. The hormones that we are administering are not a treatment but are typically used in context of routine care.
- Obese Nondiabetic Subjects: N=9 nondiabetic with BMI 24.5-29.5 kg/m2 subjects 19-45 years of age and in general good health, taking no medications, with normal glucose tolerance and no family history of diabetes. These subjects will be similar in age, ethnicity and BMI with the Type 2 Diabetes Mellitus group, and will be recruited through various means of community outreach, including notices in shops and newspapers. Will undergo pancreatic clamp
  Pancreatic Clamp: We are not performing any interventions; we are only characterizing participants using tests. The hormones that we are administering are not a treatment but are typically used in context of routine care.
Period: Overall Study
Arm/Group | Lean Diabetes Subjects | Type 2 Diabetes Mellitus Subjects | Type 1 Diabetes Mellitus Subjects | Lean Nondiabetic Subjects | Obese Nondiabetic Subjects
Started | 20 | 13 | 15 | 16 | 9
Completed | 20 | 13 | 15 | 16 | 9
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lean Diabetes Subjects | Type 2 Diabetes Mellitus Subjects | Type 1 Diabetes Mellitus Subjects | Lean Nondiabetic Subjects | Obese Nondiabetic Subjects | Total
Number analyzed (Participants) | 20 | 13 | 15 | 16 | 9 | 73
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41.5 [36.0 to 42.0] | 36.2 [32.0 to 41.0] | 28.0 [25.0 to 34.] | 26.0 [24.5 to 37.0] | 41.0 [40.0 to 41.0] | 33.5 [24.5 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 20 | 13 | 15 | 16 | 9 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 13 | 15 | 16 | 9 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race: for consistency, all subjects will be South Indian
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 20 | 13 | 15 | 16 | 9 | 73
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 20 | 13 | 15 | 16 | 9 | 73
BMI [Mean (Standard Deviation); unit: kg/m^2] | 18.3 (0.2) | 26.0 (0.3) | 20.5 (0.4) | 19.1 (0.6) | 25.4 (0.35) | 22.1 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Endogenous Glucose Production
Description: Measurements of Endogenous glucose production in each group during the low phase of the pancreatic clamp study.
Time Frame: 120 min to 240 min
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Lean Diabetes Subjects | Type 2 Diabetes Mellitus Subjects | Type 1 Diabetes Mellitus Subjects | Lean Nondiabetic Subjects | Obese Nondiabetic Subjects
Number analyzed (Participants) | 20 | 13 | 15 | 16 | 9
mg/kg/min | 0.5 (0.1) | 0.84 (0.1) | 0.6 (0.1) | 0.4 (0.1) | 0.7 (0.1)

2. Primary Outcome: Rate of Glucose Disposal (RD).
Description: Peripheral Insulin Sensitivity (RD) measured by the change in Glucose Rates of Disappearance in each group during the low phase of the pancreatic clamp study.
Time Frame: 240 min to 360 min
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Lean Diabetes Subjects | Type 2 Diabetes Mellitus Subjects | Type 1 Diabetes Mellitus Subjects | Lean Nondiabetic Subjects | Obese Nondiabetic Subjects
Number analyzed (Participants) | 20 | 13 | 15 | 16 | 9
mg/kg/min | 10.1 (0.7) | 4.2 (0.5) | 8.5 (0.4) | 10.8 (0.7) | 7.6 (0.5)

3. Secondary Outcome: Insulin Secretion
Description: Insulin secretion assessed during a 120min mixed-meal tolerance test (MMTT). Insulin secretion was calculated from the C-peptide deconvolution studies with measurements mg/kg/min using the trapezoidal method.
Time Frame: 0 min to 120 min
Measure: Median (Inter-Quartile Range); unit: mg/kg/min
Arm/Group | Lean Diabetes Subjects | Type 2 Diabetes Mellitus Subjects | Type 1 Diabetes Mellitus Subjects | Lean Nondiabetic Subjects | Obese Nondiabetic Subjects
Number analyzed (Participants) | 20 | 13 | 15 | 16 | 9
mg/kg/min | 383.0 [199.8 to 557.3] | 839.5 [609.8 to 1366.6] | 0.09 [0.09 to 0.09] | 591.1 [547.1 to 1260.5] | 1277.0 [1109.0 to 1599.1]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 month.
Arm/Group | Type 2 Diabetes Mellitus Subjects | Lean Diabetes Subjects | Type 1 Diabetes Mellitus Subjects | Lean Nondiabetic Subjects | Obese Nondiabetic Subjects
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/20 | 0/15 | 0/16 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/20 | 0/15 | 0/16 | 0/9
Other Adverse Events (participants affected / at risk) | 0/13 | 0/20 | 0/15 | 0/16 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT02987335/Prot_SAP_000.pdf